CLINICAL TRIAL: NCT02870998
Title: Comparing the Impacts of Two Versions of a Continuing Education Activity Targeted at COPD Case Managers on Educational Outcomes
Brief Title: Impacts of a Continuing Education Activity Targeted at COPD Case Managers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Louis-Philippe Boulet, MD, Laval University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MP-10-2016-2591
Record Dates: First submitted 2016-03-15; First posted 2016-08-18 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Lung Diseases, Obstructive
MeSH Terms: conditions — Lung Diseases, Obstructive | interventions — Supervised Machine Learning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active learning (Experimental): Educational strategies will be used to foster active learning.
  Interventions: Other: Active learning
- Passive learning (Active Comparator): Traditional educational strategies (lecture) will be used.
  Interventions: Other: Passive learning

INTERVENTIONS:
Other: Active learning — 1-day continuing education activity consisting of a lecture on patient education.
  Arms: Active learning
Other: Passive learning — 1-day continuing education activity consisting of a brief lecture on patient education and workshops.
  Arms: Passive learning

SUMMARY:
This study aims to compare the impacts of two versions of a continuing education activity targeted at COPD case managers on educational outcomes: 1) participation; 2) satisfaction; 3) learning; 4) competence; 5) performance; 6) patient health outcomes.

DETAILED DESCRIPTION:
This study has a quasi-experimental design. The study is based on the Expanded Outcomes Framework for Planning and Assessing Continung Medical Education by Moore (2009). One groupe of participants will attend the former version of the continuing education activity, and the other group will attend its new version.

Data will be collected at T0 (before the activity, which will be held at T1); at T2 (immediately after the activity); at T3 (1-month post-activity); at T4 (2-month post-activity); at T5 (4-month post-activity); at T6 (10-month post-activity).

Participation will be assessed at T0. Satisfaction will be assessed at T2. Learning will be assessed at T0 and T3. Competence will be assessed at T2. Performance will be assessed at T4. Patient health outcomes will be assessed at T5 and T6.

ELIGIBILITY:
Inclusion criteria for attendees:

* Attending the continuing education activity
* Providing patient education to individuals with COPD in professional setting.

Exclusion criteria for attendees:

* None

Inclusion criteria for COPD patients:

* Doctor-diagnosed COPD.

Exclusion criteria for attendees:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Performance | 2-month post-intervention
  We will videotape patient education intervention delivered by attendees in their professional practice and will assess the quality of the delivered patient education intervention using a set a pre-defined criteria.

SECONDARY OUTCOMES:
Satisfaction | Immediately post-intervention
  We will measured the extent to which attendees' expectations about the continuing education activity are met, using a self-administered questionnaire.
Learning | Prior to and 1-month post-intervention
  We will measured declarative and procedural knowledge about patient education in attendees, using a validated self-administered questionnaire.
Competence | Prior and immediately post-intervention
  We will measure attendees' self-reported competences in achieving learning activity objectives, using a self-administered questionnaire.
Patient health outcomes | 4-month and 10-month post-intervention
  We will measured COPD patients' health-related quality of life, self-management skills, and health utilization, using validated interviewer-administered questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The datasets during and/or analysed during the current study will be available from the principal investigator on reasonable request.

REFERENCES:
- [Derived] Gagne M, Lauzier S, Babineau-Therrien J, Hamel C, Penney SE, Bourbeau J, Moisan J, Boulet LP. COPD-Specific Self-Management Support Provided by Trained Educators in Everyday Practice is Associated with Improved Quality of Life, Health-Directed Behaviors, and Skill and Technique Acquisition: A Convergent Embedded Mixed-Methods Study. Patient. 2020 Feb;13(1):103-119. doi: 10.1007/s40271-019-00386-7. PMID 31502238
- [Derived] Gagne M, Moisan J, Lauzier S, Hamel C, Cote P, Bourbeau J, Boulet LP. Comparative impact of two continuing education activities targeted at COPD educators on educational outcomes: protocol for a non-randomized controlled study using mixed methods. BMC Health Serv Res. 2018 Jun 18;18(1):460. doi: 10.1186/s12913-018-3284-6. PMID 29914484

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT02870998/Prot_SAP_000.pdf